CLINICAL TRIAL: NCT00002737
Title: A RANDOMIZED PHASE II TRIAL OF INTERFERON ALPHA-2A WITH AND WITHOUT 13-CIS RETINOIC ACID IN PATIENTS WITH PROGRESSIVE MEASURABLE METASTATIC RENAL CELL CARCINOMA. Amendment Protocol: Extension to a Randomized Phase III Trial
Brief Title: Interferon Alfa With or Without Isotretinoin in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30951; EORTC-30951
Record Dates: First submitted 1999-11-01; First posted 2004-05-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; Drug Therapy; Isotretinoin

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: chemotherapy
Drug: isotretinoin

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of the cancer cells and slow the growth of kidney cancer. Isotretinoin may help kidney cancer cells develop into normal cells. It is not yet known whether interferon alfa plus isotretinoin is more effective than interferon alfa alone for kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with or without isotretinoin in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate and response duration of interferon alfa with vs without isotretinoin in patients with bidimensionally measurable progressive metastases from renal cell cancer. II. Assess the toxic effects of these regimens in this patients population. III. Determine the overall survival of this patient population treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of two treatment arms. Arm I: Patients receive interferon alfa subcutaneously daily. Arm II: Patients receive interferon alfa as in arm I plus oral isotretinoin daily. Treatment continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients are followed until death.

PROJECTED ACCRUAL: A total of 296 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic renal cell adenocarcinoma Histologic confirmation of metastases desirable Progression of metastases within 2 months of study No clinically manifest CNS metastasis Bidimensionally measurable metastases, as follows: Lung lesion with diameter greater than 2 cm Superficial lymph node or skin or subcutaneous lesion with diameter greater than 2.5 cm Lymph node in the mediastinum or retroperitoneal region, liver lesion, or soft tissue lesion visible on CT or ultrasound with initial diameter greater than 2.5 cm No bone lesion without surrounding, measurable soft tissue lesion

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0 or 1 Life expectancy: At least 90 days Hematopoietic: WBC greater than 3,000/mm3 OR Absolute granulocyte count greater than 1,500/mm3 OR Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.1 mg/dL Lipids no greater than 1.5 times normal Renal: Creatinine no greater than 1.6 mg/dL Cardiovascular: No congestive heart failure No significant arrhythmia No complete bundle branch block Pulmonary: No serious concurrent pulmonary illness Other: No recent uncontrolled bleeding No serous effusion No history of autoimmune disease No controlled or uncontrolled active infection No seizure disorder or compromised CNS function No secondary gastrointestinal dysfunction that could interfere with drug absorption No psychological condition that would preclude participation or consent No second malignancy except basal cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: At least 3 months since irradiation of target lesions Subsequent progression or new lesion required No concurrent radiotherapy Surgery: Prior nephrectomy required No concurrent surgery Other: No concurrent tetracyclines or hepatotoxic drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 1996-03; Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Aass, MD, Study Chair — Norwegian Radium Hospital
Locations (27):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- National Institute of Oncology, Budapest, Hungary
- Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- Netherlands (8):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Norwegian Radium Hospital, Oslo, Norway
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- Switzerland (7):
  - Kantonspital Aarau, Aarau
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Ratisches Kantons und Regionalspital, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - Saint Gallen, Sankt Gallen
  - Universitaetsspital, Zurich
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Bristol Royal Infirmary, Bristol, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Result] Aass N, De Mulder PH, Mickisch GH, Mulders P, van Oosterom AT, van Poppel H, Fossa SD, de Prijck L, Sylvester RJ. Randomized phase II/III trial of interferon Alfa-2a with and without 13-cis-retinoic acid in patients with progressive metastatic renal cell Carcinoma: the European Organisation for Research and Treatment of Cancer Genito-Urinary Tract Cancer Group (EORTC 30951). J Clin Oncol. 2005 Jun 20;23(18):4172-8. doi: 10.1200/JCO.2005.07.114. PMID 15961764